CLINICAL TRIAL: NCT05956782
Title: A Dyad-based Multiple Behavior Intervention for Reducing Lung Cancer Symptoms - a Pilot Randomized Control Trial (Breathe Easier II)
Brief Title: Breathe Easier II: A Dyad-based Multiple Behavior Intervention
Acronym: BE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Brown University (Other)
Responsible Party: Principal Investigator, Karen Kane McDonnell, Associate Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00112653
Record Dates: First submitted 2023-05-19; First posted 2023-07-21 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Lung Cancer, Nonsmall Cell; COPD; Self-Management; Physical Inactivity; Stress; Quality of Life
Keywords: Cancer Survivorship
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pulmonary Disease, Chronic Obstructive; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: A 6-month, two-group, longitudinal pilot RCT study with a pre- and post-test design. The intervention is 12 weeks followed by a 12 week taper. Two groups include an intervention group and an attention control group.
Who Masked: Outcomes Assessor
Masking Description: One staff person who is the outcome assessor will be blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention Control (Active Comparator): 1. Education: Each survivor will receive a copy of "Facing Forward; Life After Cancer Treatment" (No. 18-2424, March 2018). Each family member or friend will receive "When Someone You Love is Being Treated for Cancer" (No. 14-5726, May 2014). Specific parts of booklets will be reviewed during the 15-minute/per participant telephone "chat".
  2. Telephone "Chats": The primary purpose is study retention. After the first 12-week period ends the weekly chats will be tapered for 12 weeks.
  3. One text message delivered weekly by telephone is a reminder of the day and time of the chat(s).
  Tobacco Use Reduction: Many survivors of lung cancer struggle with nicotine addiction; smoking cessation and relapse prevention content will be made available to current smokers (The FOREVER FREE program - a free, twelve short booklet evidence-based resource created by the H. Lee Moffitt Cancer Center & Research Institute at the University of South Florida).
  Interventions: Behavioral: Breathe Easier
- BE Intervention Group (Experimental): 1. The BE Manual is an educational resource for Managing Stress, Increasing Physical Activity (PA) and Stopping Smoking and Staying Smoke free.
  2. A timed, weekly telephone counseling session (60 min./dyad max) will be recorded. The purpose is to provide social support with SMART goal setting, adherence monitoring, encouragement..
  3. Breathing Exercises and Meditations are incorporated into the BE Manual and sent by a link via text messages.
  4. A Texting Library provides additional education, support, and encouragement daily. There are 5 story lines: BE Active, BE Kind to Yourself, BE Supportive and BE Smoke free (offered to current smokers only). Stay Smoke free will be instituted once tobacco use has stopped.
  5. Weekly Logs for tracking goals and progress with behavior changes (PA, breathing practices and meditations) and a pedometer are provided. After 12 weeks, the calls and texts will be tapered.
  Interventions: Behavioral: Breathe Easier

INTERVENTIONS:
Behavioral: Breathe Easier — See Intervention Group (IG) description.

SUMMARY:
This pilot randomized control trial (RCT) will test a 12-week, multiple behavior intervention physical activity and stress management for survivors with early stage lung cancer (stages I-III) and their family members (1 survivor + 1 family member or friend = 1 dyad). The long-term goal of this research is to improve health outcomes for survivors of lung cancer and their family members.

The goals of the intervention, Breathe Easier, are symptom reduction (less breathlessness, less fatigue, less stress) and change in multiple behaviors (increase in stress management and increase in physical activity, and decrease tobacco use - if appropriate).

Our aim is: To conduct a 6-month, two-group, pilot randomized control trial intervention study with a pre- and post-test study design to estimate preliminary intervention effects on (a) reduction of symptoms (breathlessness, fatigue, and stress) in survivors of non small cell lung cancer (stages I-III) and family members or friends; (b) increase in physical activity behaviors immediately following the intervention and at 3-months; (c) increase in stress management strategies immediately following the intervention and at 3-months; (d) reduction in smoking behavior among participants who smoke tobacco products at study entry immediately following the intervention at 3-months.

DETAILED DESCRIPTION:
Lung cancer is the second most diagnosed malignancy and the leading cause of cancer deaths, accounting for more annual deaths than breast, prostate, and colorectal cancer combined. Approximately 80% will be diagnosed with NSCLC, and about 42.1% will present with early-stage or localized disease (stages I-III). Improvements in screening and treatment have led to better outcomes for early-stage diagnoses. As early detection improves along with treatments, the current 5-year survival rates (57%, stages I-III; 70%, stage I) are projected to improve.

Only a small percentage (5-10%) of patients with lung cancer are asymptomatic at diagnosis. Cough, dyspnea, chest discomfort, and fatigue are common symptoms. Up to 80% of long-term lung cancer survivors report smoking-related comorbidities such as chronic obstructive pulmonary disease (COPD) and heart disease. Thoracic surgery, radiation and chemotherapy may improve or worsen symptoms. After curative surgery, survivors describe persistent physical and psychological symptoms negatively affecting their QOL. The extent of the resection, co-morbid conditions, and smoking status further exacerbate symptoms. Symptoms may be intensified by smoking or withdrawal from tobacco. Nicotine withdrawal brings about a variety of physical and psychological symptoms that can temporarily intensify the symptom burden. Overall, survivors with lung cancer experience more symptom distress than survivors with other types of cancer.

Multiple unhealthy behaviors often accompany smoking, including lower physical activity levels and ineffective stress-management skills. Researchers have examined the prevalence of multiple health behaviors in lung cancer survivors; four studies targeted dyads. In one cross-sectional study data from 37 dyads (mostly white, non-Hispanic) showed high rates of smoking (43%, survivors; 30%, family members (FMs)) and physical inactivity (84%, each group). In terms of readiness to change, within 6 months post-diagnosis, 63% of patients and 81% of FMs were ready to increase their physical activity, and 88% of patients and 91% of FMs were prepared to stop smoking. A qualitative study involving 26 African American dyads, within 7 years post-diagnosis, revealed fewer current smokers (15%, survivors; 8% FMs) and persistent physical inactivity (65% survivors; 42% FMs). Two more recent studies collected similar data from survivors and their caregivers (mostly white, non-Hispanic) within 1-month post-diagnosis and 6-months post thoracic surgery reported that survivors and caregivers were receptive to educational and lifestyle behavior modification programs.

Evidence strongly suggests that smoking cessation and physical exercise interventions (individually administered) improve QOL and other outcomes; furthermore, exercise therapy is a well-tolerated, safe, and feasible adjunct therapy that can mitigate several diseases- and treatment-related side effects. Mounting evidence suggests that survivors with early-stage lung cancer benefit from regular physical activity. In a study of 175 long-term lung cancer survivors, the 27% who reported meeting physical activity guidelines also reported a higher QOL. Two pilot studies provided "proof of principle" and showed aerobic training (continuous activity involving large muscle groups) is safe and feasible for survivors of early-stage lung cancer. Thus, it is hoped that this research will advance scientific knowledge about these behaviors being complementary and producing a synergistic effect on behavior change and symptom management.

Family, friends, and especially partners of survivors of lung cancer must cope with its physical and psychological impact on the survivor, themselves, and others. It is important to recognize that survivors and their family members react to a serious illness as a unit, and as a result they both have a genuine need for help from healthcare providers. Partners not only provide emotional and practical support, but they must also cope with their own concerns, including the uncertainty surrounding the course of the illness, fear of losing their partner and the impact of their health behaviors. More than half of the partners of lung cancer survivors report negative emotional effects of being the support person. Relationships between survivors and partners are affected by the cancer also. An emerging consensus in the literature is that when both the survivor and family member are treated simultaneously, the well-being of each individual improves. When their needs are not addressed, family members are at risk for impaired health. Interestingly, most health behavior-related interventions focus on an individual's behaviors. Yet, health behaviors tend to cluster in families and social networks. The past decade has seen a growth in interventions exploring the effects of family members (and their behaviors) on each other when a serious illness is diagnosed in one of them. A greater emphasis is needed on interventions that target families, not only the survivor.

This proposed research represents the next step toward understanding the best ways to improve multiple behaviors and therefore reduce the burden of symptoms among survivors of lung cancer and their family members. The long-term contribution of this research is to advance scientific knowledge about improving outcomes for the survivors of localized NSCLC (stages I-III) and their family members.

Theoretical Framework: Individual and family self-management theory (IFSMT) is a descriptive mid-range theory developed based on conceptual and theoretical perspectives from Systems Theory, Social Learning Theory/Social Cognitive Theory, and Social Support Theory and research related to self-management (SM) of chronic illnesses. IFSMT proposes that successful change in the self-management of behaviors (physical inactivity and stress management) after a diagnosis of lung cancer requires active involvement by the survivor coupled with family support. IFSMT encompasses three broad dimensions: context, process, and outcomes. The context dimension can directly impact individual and family engagement in the self-management process and, therefore, the outcomes. Within the process dimension, self-regulation is the process used to change behavior. Social support enhances the capacity to change and includes influence and collaboration among individuals and family members. In this study, the intervention impacts the self-management process by promoting self-efficacy, self-regulation, and social support; enhancing these three factors, in turn, will lead to improved proximal outcomes (increased stress management and physical activity and reduction in tobacco smoking, relapse prevention) and distal outcomes (reduction of symptoms of dyspnea, fatigue, and stress) for all participants.

Design: This study will use a 6-month, longitudinal, two-group, repeated-measures, attention control pilot RCT design.

During an enrollment period, the research team will provide information about the study, execute an informed consent process, and collect baseline data. After baseline data is collected, participants will be instructed about the wearing of a wrist accelerometer and responding to Ecological Momentary Assessment (EMA) surveys on their cell phones for a 7-day period prior to randomization. All participants will be instructed on how to keep an accelerometer log and how to respond to mobile EMA surveys. At the end of the 7-day period, accelerometers are returned and completed data is confirmed, the randomization process will take place.

The randomization strategy will be determined by the statistician. Based on a grid developed by the statistician each envelope identified by study number only will contain the identification of the study randomized condition (Breathe Easier II [intervention] or attention control.

Statistical Analysis As a preliminary step, baseline demographic characteristics and medical histories will be compared between groups (intervention and control), for survivors and family members separately, as well as aggregated across the dyads, using t-tests (for continuous variables) and chi-squared tests (for categorical variables). This is only a preliminary step, dyadic analysis follows. Additionally within-dyad correlations in baseline measures may differ across dyads. For example, whether the association between baseline sleep and physical activity within-dyad differs across pairs. A dyadic analysis will be used as follows: using a series of longitudinal mixed effects models, the effect of intervention vs. control on changes in symptoms (shortness of breath and fatigue) after baseline will be estimated. Specifically, mean symptom at follow-up (end of intervention, 3- and 6-month follow-up) will be simultaneously regressed on group, time, group x time, baseline value, and covariates not balanced by randomization. In addition, models will control for smoking status. Interactions between smoking status at study entry within the intervention group will be explored, as it is hypothesized that the effect of the intervention will be greatest among those who were smoking at study entry.

Models will include a subject-specific intercept to adjust for repeated measures of the outcome within participants. Models will be run for the study pool (survivors and family members, considered as dyadic units) with clustering by dyad. This will adjust standard errors for the dependence of outcomes within the dyad by including an interaction term between participant (survivor vs. family member) and treatment group (intervention vs. control).

As this is a pilot study, the interest is in estimating effect sizes and corresponding 95% confidence intervals, rather than strict statistical hypothesis testing. Similar analyses will be run to estimate intervention effects on physical activity behavior (exercise capacity, minutes of moderate-intensity activity both objectively measured and self-reported, and sedentary time) and to explore intervention effects on changes in exploratory variables (context and process measures) over time. Finally, using a series of longitudinal regression models implemented with generalized estimating equations with robust standard errors and clustering by dyad, the effect on smoking outcomes at follow-up (abstinence) will be estimated. Specifically, binary indicators of abstinence on treatment assigned (intervention vs. control) and potential covariates (including variables not balanced by randomization) will be regressed using binomial errors, a logit link function, and a working unstructured correlation to accommodate within-subject correlation. Coefficients will be standardized, and models run with the sub-sample of dyads where at least one member smoked at study entry. All models will be run on the intent to treat the sample with all randomized participants included. Changes over time in secondary measured variables (e.g., process measures, sleep) and potential moderators of the intervention effect, will be explored using a similar analytic strategy to that described above. Moderator analyses will be explored by including main effects of the potential moderators (in the model of physical activity behavior for example), as well as the interaction with the treatment group.

ELIGIBILITY:
Vulnerable populations: Three groups (prisoners, pregnant women and unborn fetuses, and children) will not be included in this study because there may be unknown risks. Prisoners will be excluded because if a survivor or a family member were a current prisoner, it would be impractical to expect an individual to fully participate for 6 months.

Pregnant women and unborn fetuses will be excluded because there may be unknown risks.

Inclusion of adolescents and children: Adolescents and children will be excluded also because they are younger than the Inclusion Criteria requirement of 21 years of age. Strategies to obtain representation of children in this study would not be appropriate, as they do not get the disease. Also, they will be excluded from participating as family members.

Table 3. Inclusion and Exclusion Criteria

Inclusion Criteria: Survivors

* Completed primary treatment for localized NSCLC (stages I-III). Survivors receiving adjuvant therapy are eligible.
* Willing to use a cell phone capable of receiving text messages
* Willing to complete a 12-week, home-based intervention program that includes face-to-face and telephone interaction
* Willing to consider behavior change at this time
* A family member or friend is willing to participate who is at least 21 years old
* Able to speak and read English
* Capable of informed consent
* A health clearance form is signed by a health care provider prior to enrollment

Inclusion Criteria: Family Members or Friends

* Willing to use a cell phone capable of receiving text messages
* Willing to complete a 12-week, home-based intervention program that includes face-to-face and telephone interaction
* Willing to consider behavior change at this time
* Has an eligible family member willing to participate who is at least 21 years old
* Able to speak and read English
* Capable of informed consent
* A health clearance form signed by a health care provider prior to enrollment

Exclusion Criteria: Both

* A known diagnosis of advanced lung cancer (stage IV)
* Physical activity is not recommended
* A history of recurrent falls
* A substantial mobility impairment related to rheumatoid arthritis, cerebral palsy, muscular dystrophy, multiple sclerosis, paralysis, Parkinson's disease, stroke

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Physical function behavior change | Daily for 6 months
  Measured by self-reported step counting using a pedometer and documented on a daily log.
Physical function behavior change | Pre-intervention (Baseline) and post 3-months
  Objectively measured by wearing an Accelerometer (on the participant's wrist with a velcro band) for 7 days. Measures physical activity intensity (sedentary, light, moderate, vigorous, and very vigorous).
Physical function behavior change | Pre-intervention (Baseline) and post 6-months
  Objectively measured by wearing an Accelerometer (on the participant's wrist with a velcro band) for 7 days. Measures physical activity intensity (sedentary, light, moderate, vigorous, and very vigorous).
Physical function behavior change | Pre-intervention (Baseline) and post 3-months
  Objectively measured by a Six-minutes Walk Test.
  Specifically measures physical activity/exercise tolerance. Score = distance traveled in 6 min. measured in meters.
Physical function behavior change | Pre-intervention (Baseline) and post 6-months
  Objectively measured by a Six-minutes Walk Test.
  Specifically measures physical activity/exercise tolerance. Score = distance traveled in 6 min. measured in meters.
Stress management behavior change | Daily for 6 months
  Measured by self-reported practice of breathing exercises documented on daily logs.
Stress management behavior change | Daily for 6 months
  Measured by self-reported meditation practice documented on daily logs.
Change in the symptom of dyspnea | Pre-intervention (Baseline) and post 3-months
  As measured by a validated instrument:
  Functional Assessment of Chronic Illness Therapy (FACIT)-Dyspnea Short Form (Part 1)
  Measured by 10 items with a 4-point rating scale measuring shortness of breath (SOB) over the past 7 days (0 = not SOB; 1 = mildly SOB; 2= moderately SOB; 3 = severe SOB). Total score range 0 to 40. The higher the score measures worse SOB.
Change in the symptom of dyspnea | Pre-intervention (Baseline) and post 6-months
  As measured by a validated instrument:
  Functional Assessment of Chronic Illness Therapy (FACIT)-Dyspnea Short Form (Part 1)
  Measured by 10 items with a 4-point rating scale measuring shortness of breath (SOB) over the past 7 days (0 = not SOB; 1 = mildly SOB; 2= moderately SOB; 3 = severe SOB). Total score range 0 to 40. The higher the score measures worse SOB.
Change in the symptom of dyspnea | Pre-intervention (Baseline) and post 3-months
  As measured by a validated instrument:
  Functional Assessment of Chronic Illness Therapy (FACIT)-Dyspnea Short Form (Part 2).
  Measured by 10 items with a 4-point rating scale measuring functional limitations due to shortness of breath (SOB) over the past 7 days (0 = no difficulty, 1 = little difficulty; 2= some difficulty; 3 = much difficulty). Total score range 0 to 40. The higher the score measures greater functional difficulty due to SOB.
Change in the symptom of dyspnea | Pre-intervention (Baseline) and post 6-months
  As measured by a validated instrument:
  Functional Assessment of Chronic Illness Therapy (FACIT)-Dyspnea Short Form (Part 2).
  Measured by 10 items with a 4-point rating scale measuring functional limitations due to shortness of breath (SOB) over the past 7 days (0 = no difficulty, 1 = little difficulty; 2= some difficulty; 3 = much difficulty). Total score range 0 to 40. The higher the score measures greater functional difficulty due to SOB.
Change in the symptom of breathlessness | Pre-intervention (Baseline) and post 3-months
  As measured by validated instrument:
  Modified Medical Research Council - Dyspnea (mMRC) measures respiratory disability.
  1 item measures perceived breathlessness. There are 5 statements describing respiratory disability. Scores range from 1 to 5. No disability = "I only get breathless with strenuous exercise" (Grade 1) to "I am too breathless to leave the house" (Grade 5). The higher the score the greater the disability.
Change in the symptom of breathlessness | Pre-intervention (Baseline) and post 6-months
  As measured by validated instrument:
  Modified Medical Research Council - Dyspnea (mMRC) measures respiratory disability.
  1 item measures perceived breathlessness. There are 5 statements describing respiratory disability. Scores range from 1 to 5. No disability = "I only get breathless with strenuous exercise" (Grade 1) to "I am too breathless to leave the house" (Grade 5). The higher the score the greater the disability.
Change in the symptom of fatigue | Pre-intervention (Baseline) and post 3-months
  As measured by a validated instrument:
  Functional Assessment of Chronic Illness Therapy Scale (FACIT)-Fatigue (V.4) measures fatigue.
  Measured by 13-items with a 4-point rating scale (4 = not fatigued at all; 0 = very much fatigued). Score range is 6 to 52. The higher the score the less fatigue.
Change in the symptom of fatigue | Pre-intervention (Baseline) and post 6-months
  As measured by a validated instrument:
  Functional Assessment of Chronic Illness Therapy Scale (FACIT)-Fatigue (V.4) measures fatigue.
  Measured by 13-items with a 4-point rating scale (4 = not fatigued at all; 0 = very much fatigued). Score range is 6 to 52. The higher the score the less fatigue.
Change in perceived stress | Pre-intervention (Baseline) and post 3-months
  As measured by a validated instrument:
  Perceived Stress Scale measures perceived stress using a 10-item scale. There are 5 response items (0 = never, 1 = almost never, 2 = sometimes, 3 = fairly often, 4 = very often). Score ranges from 0 to 40. The higher the score the greater perceived stress.
Change in perceived stress | Pre-intervention (Baseline) and post 6-months
  As measured by a validated instrument:
  Perceived Stress Scale measures perceived stress using a 10-item scale. There are 5 response items (0 = never, 1 = almost never, 2 = sometimes, 3 = fairly often, 4 = very often). Score ranges from 0 to 40. The higher the score the greater perceived stress.

SECONDARY OUTCOMES:
Tobacco use abstinence | Pre-intervention (Baseline) and post 3-months
  Abstinence since quit date (score options yes/no)
Tobacco use abstinence | Pre-intervention (Baseline) and post 6-months
  Abstinence since quit date (score options yes/no)
Tobacco use abstinence | Pre-intervention (Baseline) and post 3-month
  Number of days without smoking in previous 7 days (score options: 0 to 7 days) will be measured by self report. The greater the number the greater daily abstinence.
Tobacco use abstinence | Pre-intervention (Baseline) and post 6-months
  Number of days without smoking in previous 7 days (score options: 0 to 7 days) will be measured by self report. The greater the number the greater daily abstinence.
Tobacco use abstinence | Pre-intervention (Baseline) and post 3-months
  Saliva cotinine analysis: immune-chromatographic assay that quantifies cotinine (a major metabolite of nicotine with a relatively long half-life [10-40 hr]) will verify tobacco abstinence. Results will be reported as ___ng/ml. Result interpretations will be guided by https://salimetrics.com/guidelines-for-interpreting-cotinine-levels-united-states.
Tobacco use abstinence | Pre-intervention (Baseline) and post 6-months
  Saliva cotinine analysis: immune-chromatographic assay that quantifies cotinine (a major metabolite of nicotine with a relatively long half-life [10-40 hr]) will verify tobacco abstinence. Results will be reported as ___ng/ml. Result interpretations will be guided by https://salimetrics.com/guidelines-for-interpreting-cotinine-levels-united-states.

OTHER OUTCOMES:
Sleep quality change | Daily for 7 days at Pre-intervention (Baseline) and post 3-months
  Ecological Momentary Assessments (EMA) is described as an emerging method to assess an individual's current thoughts, affect, behavior, physical states, and contextual factors as they occur in real-time and in their natural environment.The EMA application will deliver short surveys (3 to 5 daily for 7 days) by a mobile app.
  As measured by a validated instrument:
  Sleep quality will be measured by the Pittsburgh Sleep Quality Index (PSQI). The PSQI consists of a combination of Likert-type and open-ended questions. Scores for each question range from 0 to 3 with higher scores indicating more acute sleep disturbances. Scores range from 0 to 21.
Sleep quality change | Daily for 7 days at Pre-intervention (Baseline) and post 6-months
  Ecological Momentary Assessments (EMA) is described as an emerging method to assess an individual's current thoughts, affect, behavior, physical states, and contextual factors as they occur in real-time and in their natural environment.The EMA application will deliver short surveys (3 to 5 daily for 7 days) by a mobile app.
  As measured by a validated instrument:
  Sleep quality will be measured by the Pittsburgh Sleep Quality Index (PSQI). The PSQI consists of a combination of Likert-type and open-ended questions. Scores for each question range from 0 to 3 with higher scores indicating more acute sleep disturbances. Scores range from 0 to 21.
Emotional response to dyspnea change | Daily for 7 days at Pre-intervention (Baseline) and post 3-months
  Ecological Momentary Assessments (EMA) is described as an emerging method to assess an individual's current thoughts, affect, behavior, physical states, and contextual factors as they occur in real-time and in their natural environment.The EMA application will deliver short surveys (3 to 5 daily for 7 days) by a mobile app.
  As measured by validated questions from the Patient Reported Outcomes Measurement Information System (PROMIS) Dyspnea Item Bank. The Dyspnea Emotional Response Item Bank measures emotional response. Each item (7-items) response is measured on a 5-point scale (1 = not at all, 2 = A little bit, 3 = somewhat, 4 = quite a bit, 5 = very bad). Scores range between 7 and 35. The greater the score, the greater the emotional response.
Emotional response to dyspnea change | Daily for 7 days at Pre-intervention (Baseline) and post 6-months
  Ecological Momentary Assessments (EMA) is described as an emerging method to assess an individual's current thoughts, affect, behavior, physical states, and contextual factors as they occur in real-time and in their natural environment.The EMA application will deliver short surveys (3 to 5 daily for 7 days) by a mobile app.
  As measured by validated questions from the Patient Reported Outcomes Measurement Information System (PROMIS) Dyspnea Item Bank. The Dyspnea Emotional Response Item Bank measures emotional response. Each item (7-items) response is measured on a 5-point scale (1 = not at all, 2 = A little bit, 3 = somewhat, 4 = quite a bit, 5 = very bad). Scores range between 7 and 35. The greater the score, the greater the emotional response.
Affective balance change | Daily for 7 days at Pre-intervention (Baseline) and post 3-months
  Ecological Momentary Assessments (EMA) is described as an emerging method to assess an individual's current thoughts, affect, behavior, physical states, and contextual factors as they occur in real-time and in their natural environment.The EMA application will deliver short surveys (3 to 5 daily for 7 days) by a mobile app.
  Affective Balance will be measured by a validated instrument:
  The Positive and Negative Affect Schedule (PANAS) Short Form will measure mood (affective balance). PANAS is rated on a 5-point scale: (1 = very slightly or not at all; 2 = a little, 3 = moderately, 4 = quite a bit, 5 = extremely). Scores can range from 10 to 50 for both the Positive and Negative Affect, with the lower scores representing lower levels of Positive/Negative Affect and higher scores representing higher levels of Positive/Negative Affect.
Affective balance change | Daily for 7 days at Pre-intervention (Baseline) and post 6-months
  Ecological Momentary Assessments (EMA) is described as an emerging method to assess an individual's current thoughts, affect, behavior, physical states, and contextual factors as they occur in real-time and in their natural environment.The EMA application will deliver short surveys (3 to 5 daily for 7 days) by a mobile app.
  Affective Balance will be measured by a validated instrument:
  The Positive and Negative Affect Schedule (PANAS) Short Form will measure mood (affective balance). PANAS is rated on a 5-point scale: (1 = very slightly or not at all; 2 = a little, 3 = moderately, 4 = quite a bit, 5 = extremely). Scores can range from 10 to 50 for both the Positive and Negative Affect, with the lower scores representing lower levels of Positive/Negative Affect and higher scores representing higher levels of Positive/Negative Affect.
Cognition change | Daily for 7 days at Pre-intervention (Baseline) and post 3-months
  Ecological Momentary Assessments (EMA) is described as an emerging method to assess an individual's current thoughts, affect, behavior, physical states, and contextual factors as they occur in real-time and in their natural environment.The EMA application will deliver short surveys (3 to 5 daily for 7 days) by a mobile app.
  As measured by validated questions from the Patient Reported Outcomes Measurement Information System (PROMIS) Cognition Item Bank. The PROMIS Cognitive Assessment measure cognition. Each item (4 items) will be measured on a 5 point scale (1 = none of the time, 2 = a little, 3 = somewhat, 4 = a lot, 5 = cannot do by myself). Scores range from 4 to 25. The greater the score, the more cognitively challenged.
Cognition change | Daily for 7 days at Pre-intervention (Baseline) and post 6-months
  Ecological Momentary Assessments (EMA) is described as an emerging method to assess an individual's current thoughts, affect, behavior, physical states, and contextual factors as they occur in real-time and in their natural environment.The EMA application will deliver short surveys (3 to 5 daily for 7 days) by a mobile app.
  As measured by validated questions from the Patient Reported Outcomes Measurement Information System (PROMIS) Cognition Item Bank. The PROMIS Cognitive Assessment measure cognition. Each item (4 items) will be measured on a 5 point scale (1 = none of the time, 2 = a little, 3 = somewhat, 4 = a lot, 5 = cannot do by myself). Scores range from 4 to 25. The greater the score, the more cognitively challenged.
Fatigue change | Daily for 7 days at Pre-intervention (Baseline) and post 3-months
  Ecological Momentary Assessments (EMA) is described as an emerging method to assess an individual's current thoughts, affect, behavior, physical states, and contextual factors as they occur in real-time and in their natural environment.The EMA application will deliver the same short surveys (3 to 5 daily for 7 days) by a mobile app.
  As measured by validated questions from the Patient Reported Outcomes Measurement Information System PROMIS-Ca Bank v1.0-Fatigue. 11-items measure fatigue using a 5-point scale (1 = never, 2 = rarely, 3 = sometimes, 4 = often, 5 = always). Scores range from 5 to 55. The greater the score, the greater the fatigue.
Fatigue change | Daily for 7 days at Pre-intervention (Baseline) and post 6-months
  Ecological Momentary Assessments (EMA) is described as an emerging method to assess an individual's current thoughts, affect, behavior, physical states, and contextual factors as they occur in real-time and in their natural environment.The EMA application will deliver the same short surveys (3 to 5 daily for 7 days) by a mobile app.
  As measured by validated questions from the Patient Reported Outcomes Measurement Information System PROMIS-Ca Bank v1.0-Fatigue. 11-items measure fatigue using a 5-point scale (1 = never, 2 = rarely, 3 = sometimes, 4 = often, 5 = always). Scores range from 5 to 55. The greater the score, the greater the fatigue.
Neuropathy change | Daily for 7 days at Pre-intervention (Baseline) and post 3-months
  Ecological Momentary Assessments (EMA) is described as an emerging method to assess an individual's current thoughts, affect, behavior, physical states, and contextual factors as they occur in real-time and in their natural environment.The EMA application will deliver short surveys (3 to 5 daily for 7 days) by a mobile app.
  As measured by validated questions from the Patient Reported Outcomes Measurement Information System (PROMIS). Lower extremity neuropathy will be measured by the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT/GOG-NTX-13 [Version 4]). 3- items measure neuropathy on a 5-point scale (0 = not at all, 1 = a little bit, 2 = somewhat, 3 = quite a bit, 4 = very much). Scores range from 0 to 12. Some item scores are reversed. Items are summed. The sum is multiplied by the number of items. Greater the score, the greater quality of life in relation to neuropathy.
Neuropathy change | Daily for 7 days at Pre-intervention (Baseline) and post 6-months
  Ecological Momentary Assessments (EMA) is described as an emerging method to assess an individual's current thoughts, affect, behavior, physical states, and contextual factors as they occur in real-time and in their natural environment.The EMA application will deliver short surveys (3 to 5 daily for 7 days) by a mobile app.
  As measured by validated questions from the Patient Reported Outcomes Measurement Information System (PROMIS). Lower extremity neuropathy will be measured by the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT/GOG-NTX-13 [Version 4]). 3- items measure neuropathy on a 5-point scale (0 = not at all, 1 = a little bit, 2 = somewhat, 3 = quite a bit, 4 = very much). Scores range from 0 to 12. Some item scores are reversed. Items are summed. The sum is multiplied by the number of items. Greater the score, the greater quality of life in relation to neuropathy.
Sedentary behavior change | Daily for 7 days at Pre-intervention (Baseline) and post 3-months
  Ecological Momentary Assessments (EMA) is described as an emerging method to assess an individual's current thoughts, affect, behavior, physical states, and contextual factors as they occur in real-time and in their natural environment.The EMA application will deliver the same short surveys (3 to 5 daily for 7 days) by a mobile app.
  As measured by a validated instrument:
  The Sedentary Behavior Questionnaire (SBQ) will measure sedentary behavior using an 8-item measure using a 9-response options. (0) none, (1) 15 min. or less, (2) 30 min. or less, (3) 1 hr. (4) 2 hrs., (5) 3 hrs., (6) 4 hrs., (7) 5 hrs., (8) 6 hrs. or more. Scores range from 0 to 64. The greater the score, the greater the sedentary behavior.
Sedentary behavior change | Daily for 7 days at Pre-intervention (Baseline) and post 6-months
  Ecological Momentary Assessments (EMA) is described as an emerging method to assess an individual's current thoughts, affect, behavior, physical states, and contextual factors as they occur in real-time and in their natural environment.The EMA application will deliver the same short surveys (3 to 5 daily for 7 days) by a mobile app.
  As measured by a validated instrument:
  The Sedentary Behavior Questionnaire (SBQ) will measure sedentary behavior using an 8-item measure using a 9-response options. (0) none, (1) 15 min. or less, (2) 30 min. or less, (3) 1 hr. (4) 2 hrs., (5) 3 hrs., (6) 4 hrs., (7) 5 hrs., (8) 6 hrs. or more. Scores range from 0 to 64. The greater the score, the greater the sedentary behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Karen K McDonnell, PhD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
On request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Protocol will be submitted for publication in 2024. Data will be shared post statistical analysis by publication in open access journal.
Access Criteria: Undecided

REFERENCES:
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer statistics, 2022. CA Cancer J Clin. 2022 Jan;72(1):7-33. doi: 10.3322/caac.21708. Epub 2022 Jan 12. PMID 35020204
- [Background] Cox-Martin E, Cox MG, Basen-Engquist K, Bradley C, Blalock JA. Changing multiple health behaviors in cancer survivors: smoking and exercise. Psychol Health Med. 2020 Mar;25(3):331-343. doi: 10.1080/13548506.2019.1679849. Epub 2019 Oct 19. PMID 31630537
- [Background] Bluethmann SM, Mariotto AB, Rowland JH. Anticipating the "Silver Tsunami": Prevalence Trajectories and Comorbidity Burden among Older Cancer Survivors in the United States. Cancer Epidemiol Biomarkers Prev. 2016 Jul;25(7):1029-36. doi: 10.1158/1055-9965.EPI-16-0133. PMID 27371756
- [Background] Lemjabbar-Alaoui H, Hassan OU, Yang YW, Buchanan P. Lung cancer: Biology and treatment options. Biochim Biophys Acta. 2015 Dec;1856(2):189-210. doi: 10.1016/j.bbcan.2015.08.002. Epub 2015 Aug 19. PMID 26297204
- [Background] Young RP, Hopkins RJ, Christmas T, Black PN, Metcalf P, Gamble GD. COPD prevalence is increased in lung cancer, independent of age, sex and smoking history. Eur Respir J. 2009 Aug;34(2):380-6. doi: 10.1183/09031936.00144208. Epub 2009 Feb 5. PMID 19196816
- [Background] Celli BR. Chronic obstructive pulmonary disease and lung cancer: common pathogenesis, shared clinical challenges. Proc Am Thorac Soc. 2012 May;9(2):74-9. doi: 10.1513/pats.201107-039MS. PMID 22550249
- [Background] McDonnell KK, Bullock LF, Hollen PJ, Heath J, Kozower BD. Emerging issues on the impact of smoking on health-related quality of life in patients with lung cancer and their families. Clin J Oncol Nurs. 2014 Apr;18(2):171-81. doi: 10.1188/14.CJON.18-02AP. PMID 24534075
- [Background] Cataldo JK, Dubey S, Prochaska JJ. Smoking cessation: an integral part of lung cancer treatment. Oncology. 2010;78(5-6):289-301. doi: 10.1159/000319937. Epub 2010 Aug 11. PMID 20699622
- [Background] Lowery AE, Krebs P, Coups EJ, Feinstein MB, Burkhalter JE, Park BJ, Ostroff JS. Impact of symptom burden in post-surgical non-small cell lung cancer survivors. Support Care Cancer. 2014 Jan;22(1):173-80. doi: 10.1007/s00520-013-1968-3. Epub 2013 Sep 10. PMID 24018910
- [Background] Vijayvergia N, Shah PC, Denlinger CS. Survivorship in Non-Small Cell Lung Cancer: Challenges Faced and Steps Forward. J Natl Compr Canc Netw. 2015 Sep;13(9):1151-61. doi: 10.6004/jnccn.2015.0140. PMID 26358799
- [Background] Cooley ME, Finn KT, Wang Q, Roper K, Morones S, Shi L, Litrownik D, Marcoux JP, Zaner K, Hayman LL. Health behaviors, readiness to change, and interest in health promotion programs among smokers with lung cancer and their family members: a pilot study. Cancer Nurs. 2013 Mar-Apr;36(2):145-54. doi: 10.1097/NCC.0b013e31825e4359. PMID 22791213
- [Background] McDonnell KK, Owens OL, Hilfinger Messias DK, Heiney SP, Friedman DB, Campbell C, Webb LA. Health behavior changes in African American family members facing lung cancer: Tensions and compromises. Eur J Oncol Nurs. 2019 Feb;38:57-64. doi: 10.1016/j.ejon.2018.12.002. Epub 2018 Dec 7. PMID 30717937
- [Background] Roddy MK, Flores RM, Burt B, Badr H. Lifestyle behaviors and intervention preferences of early-stage lung cancer survivors and their family caregivers. Support Care Cancer. 2021 Mar;29(3):1465-1475. doi: 10.1007/s00520-020-05632-5. Epub 2020 Jul 20. PMID 32691229
- [Background] Nightingale CL, Steffen LE, Tooze JA, Petty W, Danhauer SC, Badr H, Weaver KE. Lung Cancer Patient and Caregiver Health Vulnerabilities and Interest in Health Promotion Interventions: An Exploratory Study. Glob Adv Health Med. 2019 Jul 17;8:2164956119865160. doi: 10.1177/2164956119865160. eCollection 2019. PMID 31360617
- [Background] Matulewicz RS, Sherman S, Bjurlin MA. Smoking Cessation and Cancer Survivorship. JAMA. 2020 Oct 13;324(14):1475. doi: 10.1001/jama.2020.16277. No abstract available. PMID 33048156
- [Background] Granger CL, McDonald CF, Berney S, Chao C, Denehy L. Exercise intervention to improve exercise capacity and health related quality of life for patients with Non-small cell lung cancer: a systematic review. Lung Cancer. 2011 May;72(2):139-53. doi: 10.1016/j.lungcan.2011.01.006. Epub 2011 Feb 12. PMID 21316790
- [Background] Hoffman AJ, Brintnall RA, Brown JK, Eye Av, Jones LW, Alderink G, Ritz-Holland D, Enter M, Patzelt LH, Vanotteren GM. Too sick not to exercise: using a 6-week, home-based exercise intervention for cancer-related fatigue self-management for postsurgical non-small cell lung cancer patients. Cancer Nurs. 2013 May-Jun;36(3):175-88. doi: 10.1097/NCC.0b013e31826c7763. PMID 23051872
- [Background] Jones LW, Alfano CM. Exercise-oncology research: past, present, and future. Acta Oncol. 2013 Feb;52(2):195-215. doi: 10.3109/0284186X.2012.742564. Epub 2012 Dec 17. PMID 23244677
- [Background] Paramanandam VS, Dunn V. Exercise for the management of cancer-related fatigue in lung cancer: a systematic review. Eur J Cancer Care (Engl). 2015;24(1):4-14. doi: 10.1111/ecc.12198. Epub 2014 Apr 10. PMID 24720528
- [Background] Mosher CE, Jaynes HA, Hanna N, Ostroff JS. Distressed family caregivers of lung cancer patients: an examination of psychosocial and practical challenges. Support Care Cancer. 2013 Feb;21(2):431-7. doi: 10.1007/s00520-012-1532-6. Epub 2012 Jul 14. PMID 22797839
- [Background] Mosher CE, Bakas T, Champion VL. Physical health, mental health, and life changes among family caregivers of patients with lung cancer. Oncol Nurs Forum. 2013 Jan;40(1):53-61. doi: 10.1188/13.ONF.53-61. PMID 23269770
- [Background] Siminoff LA, Wilson-Genderson M, Baker S Jr. Depressive symptoms in lung cancer patients and their family caregivers and the influence of family environment. Psychooncology. 2010 Dec;19(12):1285-93. doi: 10.1002/pon.1696. PMID 20119935
- [Background] McDonnell KK, Owens OL, Hilfinger Messias DK, Friedman DB, Newsome BR, Campbell King C, Jenerette C, Webb LA. After Ringing the Bell: Receptivity of and Preferences for Healthy Behaviors in African American Dyads Surviving Lung Cancer. Oncol Nurs Forum. 2020 May 1;47(3):281-291. doi: 10.1188/20.ONF.281-291. PMID 32301934
- [Background] Wennman-Larsen A, Persson C, Ostlund U, Wengstrom Y, Gustavsson JP. Development in quality of relationship between the significant other and the lung cancer patient as perceived by the significant other. Eur J Oncol Nurs. 2008 Dec;12(5):430-5. doi: 10.1016/j.ejon.2008.07.004. Epub 2008 Oct 8. PMID 18845476
- [Background] Badr H, Taylor CL. Effects of relationship maintenance on psychological distress and dyadic adjustment among couples coping with lung cancer. Health Psychol. 2008 Sep;27(5):616-27. doi: 10.1037/0278-6133.27.5.616. PMID 18823188
- [Background] Badr H, Krebs P. A systematic review and meta-analysis of psychosocial interventions for couples coping with cancer. Psychooncology. 2013 Aug;22(8):1688-704. doi: 10.1002/pon.3200. Epub 2012 Oct 9. PMID 23045191
- [Background] Ryan P, Sawin KJ. The Individual and Family Self-Management Theory: background and perspectives on context, process, and outcomes. Nurs Outlook. 2009 Jul-Aug;57(4):217-225.e6. doi: 10.1016/j.outlook.2008.10.004. PMID 19631064
- [Background] Chodosh J, Morton SC, Mojica W, Maglione M, Suttorp MJ, Hilton L, Rhodes S, Shekelle P. Meta-analysis: chronic disease self-management programs for older adults. Ann Intern Med. 2005 Sep 20;143(6):427-38. doi: 10.7326/0003-4819-143-6-200509200-00007. PMID 16172441
- [Background] National Cancer Institute. (2014). Facing forward: Life after cancer treatment. Bethesda, MD: National Institutes of Health.
- [Background] National Coalition of Cancer Survivorship, UCLA Cancer Survivorship Center, Oncology Nursing Society, Anthem Inc., & Genentech. (2015). Journey forward. Retrieved from http://www.journeyforward.org/about-journey-forward
- [Background] Brandon TH, Simmons VN, Sutton SK, Unrod M, Harrell PT, Meade CD, Craig BM, Lee JH, Meltzer LR. Extended Self-Help for Smoking Cessation: A Randomized Controlled Trial. Am J Prev Med. 2016 Jul;51(1):54-62. doi: 10.1016/j.amepre.2015.12.016. Epub 2016 Feb 8. PMID 26868284
- [Background] Pinto BM, Frierson GM, Rabin C, Trunzo JJ, Marcus BH. Home-based physical activity intervention for breast cancer patients. J Clin Oncol. 2005 May 20;23(15):3577-87. doi: 10.1200/JCO.2005.03.080. PMID 15908668
- [Background] Kolt GS, Schofield GM, Kerse N, Garrett N, Ashton T, Patel A. Healthy Steps trial: pedometer-based advice and physical activity for low-active older adults. Ann Fam Med. 2012 May-Jun;10(3):206-12. doi: 10.1370/afm.1345. PMID 22585884
- [Background] Van Remoortel H, Giavedoni S, Raste Y, Burtin C, Louvaris Z, Gimeno-Santos E, Langer D, Glendenning A, Hopkinson NS, Vogiatzis I, Peterson BT, Wilson F, Mann B, Rabinovich R, Puhan MA, Troosters T; PROactive consortium. Validity of activity monitors in health and chronic disease: a systematic review. Int J Behav Nutr Phys Act. 2012 Jul 9;9:84. doi: 10.1186/1479-5868-9-84. PMID 22776399
- [Background] Lehto RH, Wyatt G. Perceptions about using mindfulness therapy: a lung cancer focus group study. Cancer Nurs. 2013 Jul-Aug;36(4):E51-60. doi: 10.1097/NCC.0b013e31826d2f16. PMID 23047802
- [Background] Shennan C, Payne S, Fenlon D. What is the evidence for the use of mindfulness-based interventions in cancer care? A review. Psychooncology. 2011 Jul;20(7):681-97. doi: 10.1002/pon.1819. Epub 2010 Aug 4. PMID 20690112
- [Background] Hately J, Laurence V, Scott A, Baker R, Thomas P. Breathlessness clinics within specialist palliative care settings can improve the quality of life and functional capacity of patients with lung cancer. Palliat Med. 2003 Jul;17(5):410-7. doi: 10.1191/0269216303pm752oa. PMID 12882259
- [Background] Bonk AK. Management of dyspnea in a patient with lung cancer. Oncol Nurs Forum. 2012 May 1;39(3):257-60. doi: 10.1188/12.ONF.257-260. No abstract available. PMID 22543384
- [Background] Fiore, M. C., Jaén, C. R., Baker, T. B., Bailey, W. C., Benowitz, N. L., Curry, S. J., . . . Wewers, M. E. (2008). Clinical Practice Guideline: Treating tobacco use and dependence; 2008 update. Rockville, MD: U.S. Department of Health and Human Services, Public Health Service.
- [Background] McDonnell KK, Bullock LF, Kozower BD, Hollen PJ, Heath J, Rovnyak V. A decision aid to improve smoking abstinence for families facing cancer. Oncol Nurs Forum. 2014 Nov 1;41(6):649-58. doi: 10.1188/14.ONF.649-658. PMID 25355020
- [Background] McDonnell KK, Gallerani DG, Newsome BR, Owens OL, Beer J, Myren-Bennett AR, Regan E, Hardin JW, Webb LA. A Prospective Pilot Study Evaluating Feasibility and Preliminary Effects of Breathe Easier: A Mindfulness-based Intervention for Survivors of Lung Cancer and Their Family Members (Dyads). Integr Cancer Ther. 2020 Jan-Dec;19:1534735420969829. doi: 10.1177/1534735420969829. PMID 33118443
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Birim O, Maat AP, Kappetein AP, van Meerbeeck JP, Damhuis RA, Bogers AJ. Validation of the Charlson comorbidity index in patients with operated primary non-small cell lung cancer. Eur J Cardiothorac Surg. 2003 Jan;23(1):30-4. doi: 10.1016/s1010-7940(02)00721-2. PMID 12493500
- [Background] Creamer M, Bell R, Failla S. Psychometric properties of the Impact of Event Scale - Revised. Behav Res Ther. 2003 Dec;41(12):1489-96. doi: 10.1016/j.brat.2003.07.010. PMID 14705607
- [Background] Dibble JL, Levine TR, Park HS. The Unidimensional Relationship Closeness Scale (URCS): reliability and validity evidence for a new measure of relationship closeness. Psychol Assess. 2012 Sep;24(3):565-72. doi: 10.1037/a0026265. Epub 2011 Nov 14. PMID 22082035
- [Background] Hughes JR, Keely JP, Niaura RS, Ossip-Klein DJ, Richmond RL, Swan GE. Measures of abstinence in clinical trials: issues and recommendations. Nicotine Tob Res. 2003 Feb;5(1):13-25. PMID 12745503
- [Background] Murray RP, Connett JE, Lauger GG, Voelker HT. Error in smoking measures: effects of intervention on relations of cotinine and carbon monoxide to self-reported smoking. The Lung Health Study Research Group. Am J Public Health. 1993 Sep;83(9):1251-7. doi: 10.2105/ajph.83.9.1251. PMID 8363000
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] Marcus BH, Selby VC, Niaura RS, Rossi JS. Self-efficacy and the stages of exercise behavior change. Res Q Exerc Sport. 1992 Mar;63(1):60-6. doi: 10.1080/02701367.1992.10607557. PMID 1574662
- [Background] Velicer WF, Diclemente CC, Rossi JS, Prochaska JO. Relapse situations and self-efficacy: an integrative model. Addict Behav. 1990;15(3):271-83. doi: 10.1016/0306-4603(90)90070-e. PMID 2378287
- [Background] Zimet GD, Powell SS, Farley GK, Werkman S, Berkoff KA. Psychometric characteristics of the Multidimensional Scale of Perceived Social Support. J Pers Assess. 1990 Winter;55(3-4):610-7. doi: 10.1080/00223891.1990.9674095. PMID 2280326
- [Background] Kendzierski, D., & DeCarlo, K. J. (1991). Physical Activity Enjoyment Scale: Two validation studies. Journal of Sport and Exercise Psychology, 13(1), 50-64.
- [Background] Cohen S, Lichtenstein E. Partner behaviors that support quitting smoking. J Consult Clin Psychol. 1990 Jun;58(3):304-9. doi: 10.1037//0022-006x.58.3.304. PMID 2365893
- [Background] Prochaska JO, Velicer WF, DiClemente CC, Fava J. Measuring processes of change: applications to the cessation of smoking. J Consult Clin Psychol. 1988 Aug;56(4):520-8. doi: 10.1037//0022-006x.56.4.520. No abstract available. PMID 3198809
- [Background] Enright PL. The six-minute walk test. Respir Care. 2003 Aug;48(8):783-5. PMID 12890299
- [Background] Choi SW, Victorson DE, Yount S, Anton S, Cella D. Development of a conceptual framework and calibrated item banks to measure patient-reported dyspnea severity and related functional limitations. Value Health. 2011 Mar-Apr;14(2):291-306. doi: 10.1016/j.jval.2010.06.001. PMID 21402297
- [Background] Stenton C. The MRC breathlessness scale. Occup Med (Lond). 2008 May;58(3):226-7. doi: 10.1093/occmed/kqm162. No abstract available. PMID 18441368
- [Background] Cella D, Lai JS, Chang CH, Peterman A, Slavin M. Fatigue in cancer patients compared with fatigue in the general United States population. Cancer. 2002 Jan 15;94(2):528-38. doi: 10.1002/cncr.10245. PMID 11900238
- [Background] Yellen SB, Cella DF, Webster K, Blendowski C, Kaplan E. Measuring fatigue and other anemia-related symptoms with the Functional Assessment of Cancer Therapy (FACT) measurement system. J Pain Symptom Manage. 1997 Feb;13(2):63-74. doi: 10.1016/s0885-3924(96)00274-6. PMID 9095563
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Roberti, J. W., Harrington, L. N., & Storch, E. A. (2006). Further psychometric support for the 10-item version of the Perceived Stress Scale. Journal of College Counseling, 9(2), 135-147. https://doi.org/10.1002/j.2161-1882.2006.tb00100.x
- [Background] Davenport TE, Stevens SR, Baroni K, Van Ness JM, Snell CR. Reliability and validity of Short Form 36 Version 2 to measure health perceptions in a sub-group of individuals with fatigue. Disabil Rehabil. 2011;33(25-26):2596-604. doi: 10.3109/09638288.2011.582925. Epub 2011 Jun 20. PMID 21682669
- [Background] Kampshoff CS, Verdonck-de Leeuw IM, van Oijen MG, Sprangers MA, Buffart LM. Ecological momentary assessments among patients with cancer: A scoping review. Eur J Cancer Care (Engl). 2019 May;28(3):e13095. doi: 10.1111/ecc.13095. Epub 2019 May 14. PMID 31090160
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Norweg A, Ni P, Garshick E, O'Connor G, Wilke K, Jette AM. A multidimensional computer adaptive test approach to dyspnea assessment. Arch Phys Med Rehabil. 2011 Oct;92(10):1561-9. doi: 10.1016/j.apmr.2011.05.020. PMID 21963123
- [Background] Thompson, E. R. (2007). Development and validation of an internationally reliable short-form of the positive and negative affect schedule (PANAS). Journal of Cross-Cultural Psychology, 38(2), 227-242.
- [Background] Calhoun EA, Welshman EE, Chang CH, Lurain JR, Fishman DA, Hunt TL, Cella D. Psychometric evaluation of the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (Fact/GOG-Ntx) questionnaire for patients receiving systemic chemotherapy. Int J Gynecol Cancer. 2003 Nov-Dec;13(6):741-8. doi: 10.1111/j.1525-1438.2003.13603.x. PMID 14675309
- [Background] Rosenberg DE, Norman GJ, Wagner N, Patrick K, Calfas KJ, Sallis JF. Reliability and validity of the Sedentary Behavior Questionnaire (SBQ) for adults. J Phys Act Health. 2010 Nov;7(6):697-705. doi: 10.1123/jpah.7.6.697. PMID 21088299
- [Background] Valentine TR, Weiss DM, Jones JA, Andersen BL. Construct validity of PROMIS(R) Cognitive Function in cancer patients and noncancer controls. Health Psychol. 2019 May;38(5):351-358. doi: 10.1037/hea0000693. PMID 31045417
- [Background] Cessna JM, Jim HS, Sutton SK, Asvat Y, Small BJ, Salsman JM, Zachariah B, Fishman M, Field T, Fernandez H, Perez L, Jacobsen PB. Evaluation of the psychometric properties of the PROMIS Cancer Fatigue Short Form with cancer patients. J Psychosom Res. 2016 Feb;81:9-13. doi: 10.1016/j.jpsychores.2015.12.002. Epub 2015 Dec 11. PMID 26800633
- [Background] Motzer SA, Moseley JR, Lewis FM. Recruitment and retention of families in clinical trials with longitudinal designs. West J Nurs Res. 1997 Jun;19(3):314-33. doi: 10.1177/019394599701900304. PMID 9170990
- [Background] Northouse LL, Rosset T, Phillips L, Mood D, Schafenacker A, Kershaw T. Research with families facing cancer: the challenges of accrual and retention. Res Nurs Health. 2006 Jun;29(3):199-211. doi: 10.1002/nur.20128. PMID 16676337
- [Background] Abshire DA, McDonnell KK, Donevant SB, Corbett CF, Tavakoli AS, Felder TM, Pinto BM. Pivoting Nursing Research and Scholarship During the COVID-19 Pandemic. Nurs Res. 2021 May-Jun 01;70(3):165-172. doi: 10.1097/NNR.0000000000000493. PMID 33315760
- [Background] Kenny, D. A., Kashy, D. A., & Cook, W. L. (2006). Dyadic data analysis. New York, NY: Guilford Press.
- [Background] Liang, K. Zeger, S. Longitudinal data analysis using generalized linear models. Biometrics, 1986, 73(1), 12.
- [Background] Zeger SL, Liang KY. Longitudinal data analysis for discrete and continuous outcomes. Biometrics. 1986 Mar;42(1):121-30. PMID 3719049
- [Background] R Development Core Team. (2008). R: A language and environment for statistical computing. Vienna, Austria: R Foundation for Statistical Computing. Retrieved from http://www.R-project.org
- [Background] Kraemer HC, Mintz J, Noda A, Tinklenberg J, Yesavage JA. Caution regarding the use of pilot studies to guide power calculations for study proposals. Arch Gen Psychiatry. 2006 May;63(5):484-9. doi: 10.1001/archpsyc.63.5.484. PMID 16651505
- [Background] Leon AC, Davis LL, Kraemer HC. The role and interpretation of pilot studies in clinical research. J Psychiatr Res. 2011 May;45(5):626-9. doi: 10.1016/j.jpsychires.2010.10.008. Epub 2010 Oct 28. PMID 21035130
- [Derived] McDonnell KK, Andrews JO, Yang CH, Newsome BR, Weinkle E, Davis JE, Dunsiger S. Study Protocol for the Breathe Easier Trial: A Pilot RCT of a Dyad-Based, Multiple-Behavior Intervention for Improving Physical and Emotional Health in Survivors Facing Lung Cancer. Integr Cancer Ther. 2023 Jan-Dec;22:15347354231212876. doi: 10.1177/15347354231212876. PMID 38009546